CLINICAL TRIAL: NCT01527136
Title: A Phase 1 Study to Evaluate the Safety and Pharmacokinetic Profile of CBLB502 in Patients With Advanced Cancers
Brief Title: Entolimod in Treating Patients With Locally Advanced or Metastatic Solid Tumors That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Cleveland BioLabs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 196111; NCI-2011-03565 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 196111 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2011-12-20; First posted 2012-02-06 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — CBLB502

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (entolimod) (Experimental): Patients receive entolimod IM or SC on days 1, 4, 8, and 11. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: entolimod; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: entolimod — Given IM or SC
  Other Names: CBLB502; TLR5 agonist CBLB502; toll-like receptor 5 agonist CBLB502
Other: pharmacological study — Correlative studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of entolimod in treating patients with locally advanced or metastatic solid tumors that cannot be removed by surgery. Biological therapies, such as entolimod, may stimulate the immune system in different ways and stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety, tolerability, and maximum tolerated dose (MTD) of CBLB502 (entolimod) in patients with advanced cancers.

SECONDARY OBJECTIVES:

I. To assess any preliminary evidence of efficacy with the CBLB502 in patients with advanced cancers.

II. To evaluate pharmacokinetic (PK)/pharmacodynamic (PD) profiles of CBLB502 in patients with advanced cancers.

III. To characterize the effect, if any, of intramuscular or subcutaneous CBLB502 on QTcB.

TERTIARY OBJECTIVES:

I. To correlate pre-treatment tissue expression of toll-like receptor 5 (TLR5) with clinical activity (Response Evaluation Criteria In Solid Tumors [RECIST] tumor response) and PD response (as measured by cytokine levels) of CBLB502.

OUTLINE: This is a dose-escalation study.

Patients receive entolimod intramuscularly (IM) on day 1 and subcutaneously (SC) on days 4, 8, and 11. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures, given with the understanding that the patient has the right to withdraw from the study at any time, without prejudice
* Histologically or cytologically confirmed locally advanced, inoperable or metastatic solid tumor for which no acceptable therapy exists
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy greater than 3 months
* Platelet count >= 75 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 gm/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN, regardless of the presence of liver metastases
* Creatinine =< 2 x ULN
* Left ventricular ejection fraction (LVEF) >=45% by echocardiogram (ECHO) or multi gated acquisition scan (MUGA)
* 12-Lead Electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
* QTcB interval < 470 msec at any point prior to receiving the first dose of study drug (mean of replicate values, correction per institutional standard) and no history of Torsades des Pointes or other symptomatic QTcB abnormality
* Absence of orthostatic hypotension

Exclusion Criteria:

* Male and female subjects of child-bearing potential who do not agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received
* Previous anti-cancer chemotherapy, immunotherapy or investigational agents =< 3 weeks prior to the first day of study defined treatment; palliative radiation < 2 weeks; patients who receive gamma knife radiosurgery for brain metastases are eligible if procedure was performed > 2 weeks before treated is started, is clinically stable and is not receiving corticosteroid therapy; ongoing hormonal therapies (such as, luteinizing hormone-releasing hormone [LHRH] antagonists, megestrol, anti-estrogens, or aromatase inhibitors) are allowed
* Previous treatment with a TLR5 agonist
* Patients with a known hypersensitivity to CBLB502 or to its excipients
* Presence of neutralizing antibodies to CBLB502
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes; patients with persistent regional wall abnormalities on assessment of LVEF function are not eligible
  * History of documents congestive heart failure (New York Heart Association [NYHA] functional classification III-IV) within 6 months
  * Documented cardiomyopathy
  * Diagnosed or suspected congenital QT syndrome
  * Any history of second or third degree heart block (may be eligible if currently have a pacemaker)
  * Heart rate < 50 beats/minute on pre-entry electrocardiogram
  * Uncontrolled hypertension defined as systolic blood pressure > 160 mm Hg on 3 consecutive measurements prior to study enrollment
* Active clinically serious infections defined as >= Grade 2 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
* Substance abuse, medical, psychological, or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* Known infection with human immunodeficiency virus (HIV) or hepatitis B or hepatitis C
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF]) =< 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Women who are pregnant or breast feeding
* Patients receiving chronic treatment with steroids or another immunosuppressive agent; Note: topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular) are allowed
* Uncontrolled diabetes mellitus defined as a HgbA1c > 7%
* Patients who have received chemotherapy or targeted anticancer therapy >= 3 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover a Grade 1 toxicity before starting the trial
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
MTD of entolimod | 3 weeks
  Evaluated using National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Safety of entolimod | Up to 30 days post-treatment
  Evaluated using NCI-CTCAE Version 4.0.

SECONDARY OUTCOMES:
Efficacy of entolimod in patients with advanced cancers in terms of objective response rate (ORR) and RECIST response | Up to 3 months
  ORR will be calculated as the number of patients with a confirmed complete or partial response divided by the total number of patients. Tumor response will be summarized, and the 95% confidence interval for ORR (complete response [CR] + partial response [PR]) will be presented. Evaluated using the RECIST criteria.
PK profiles of entolimod in patients with advanced cancers | Pre-dose, 2, 4, 6, 8, 24 hours, post dose for, days 1, 4, 8 and 11
PD profiles of entolimod in patients with advanced cancers | PD plasma: pre-dose, at 2, 4 and 6 hours post dose on day 1, 4, 8, 11, 15, 22, and 43

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States